CLINICAL TRIAL: NCT04055610
Title: Effects of Gait Training for Individuals With Paraplegia Using H-MEX Exoskeleton: A Pilot Study
Brief Title: Gait Training for Individuals With Paraplegia Using the H-MEX Exoskeleton
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Hyundai Motor Company (Industry)
Responsible Party: Principal Investigator, Mi Jung Kim, Professor of Dept. of Rehabilitation Medicine, Hanyang University Seoul Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Hanyang University Hospital
Record Dates: First submitted 2019-06-19; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Spinal Cord Injuries; Paraplegia
Keywords: H-MEX powered exoskeleton; Exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H-MEX (Experimental): 10 participants with paraplegia will participate in explorative gait training using H-MEX powered exoskeleton.
  Interventions: Device: Gait training using H-MEX exoskeleton

INTERVENTIONS:
Device: Gait training using H-MEX exoskeleton — Participants will train 3 times a week for 10 weeks using H-MEX powered exoskeleton.

SUMMARY:
This study evaluates the feasibility and effects of H-MEX powered exoskeleton in individuals with paraplegia as a result of spinal cord injury.

DETAILED DESCRIPTION:
Participants with paraplegia will attend gait training using H-MEX powered exoskeleton 3 times a week for 10 weeks.

The aim of this study is to assess the impact of gait training using H-MEX powered exoskeleton on walking ability, gait analysis, medical examination, body composition, functional evaluation, laboratory findings, quality of life, and subjective experience in individuals with paraplegia.

Participants will be evaluated before, during, and after training.

ELIGIBILITY:
Inclusion Criteria:

* Neurologically stable paraplegia due to traumatic or non-traumatic spinal cord injury at least 2 months since injury
* Age more than 18 years
* Body weight less than 110kg, height between 160-180cm
* Sufficient postural stability to perform level transfer
* Sufficient upper extremity strength to use a walker or crutch

Exclusion Criteria:

* Spinal instability
* Severe joint contracture in lower extremity
* Unhealed fracture in the major weight bearing bone in the lower extremity
* Skin compromise in areas of contact with the device
* Unresolved deep vein thrombosis
* Uncontrolled hypertension or hypotension
* Severe osteoporosis or osteoporotic fracture unable to gait training
* Lower extremity spasticity exceeding 3 out of 4 (Modified Ashworth Scale) in any joint
* Upper extremity functional limitation due to weakness or contracture
* Psychological or cognitive problem that may limit the participants to understand instructions by investigator
* Any other issue that may interfere with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Dropout rate | 0-14 weeks
  Percentage of participants who drop out before the end of the training period.
Number of adverse events | 0-14 weeks
  Types and number of the adverse events both serious and non-serious events during training sessions.

SECONDARY OUTCOMES:
Changes in 6 minute walking test with H-mex exoskeleton | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Distance walked over a span of 6 minutes will be examined.
Changes in timed up and go test with H-mex exoskeleton | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Time that a participants takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down will be measured.
Changes in Berg balance test with H-mex exoskeleton | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Balance will be evaluated by using Berg balance test which is 14-item test designed to assess balance (score range: 0-56, higher values represent a better outcome).
Changes in body composition | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Body composition will be assessed by using bioelectric impedence analysis.
Changes in oxygen uptake during gait training with H-mex exoskeleton | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Average and peak oxygen uptake will be measured with participants during gait training.
Changes in heart rate during gait training with H-mex exoskeleton | Initial evaluation, mid-evaluation (after 5 weeks of training), and Final evaluation (after 10 weeks of training)
  Average and peak heart rate will be measured with participants during gait training.
Changes in bone mineral density | Initial evaluation and Final evaluation (after 10 weeks of training)
  Bone mineral density will be measured at hip and spine by dual energy X-ray absorptiometry.
Changes in colonic transit time | Initial evaluation and Final evaluation (after 10 weeks of training)
  Colonic mobility will be assessed by colonic transit time.
Changes in quality of life: Short-Form 36-Item Health Survey version 2 | Initial evaluation and Final evaluation (after 10 weeks of training)
  Quality of life will be assessed by Short-Form 36-Item Health Survey version 2 (total score range: 0-100, higher values represent a better outcome).
Changes in fear for fall | Initial evaluation and Final evaluation (after 10 weeks of training)
  Fear for fall will be assessed by fall efficacy scale which is 16-item test (score range: 16-64, higher values represent a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Mi Jung Kim, MD PhD, Principal Investigator — Department of Rehabilitation medicine, Hanyang University Hospital
Locations (1):
- Hanyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HS, Park JH, Lee HS, Lee JY, Jung JW, Park SB, Hyun DJ, Park S, Yoon J, Lim H, Choi YY, Kim MJ. Effects of Wearable Powered Exoskeletal Training on Functional Mobility, Physiological Health and Quality of Life in Non-ambulatory Spinal Cord Injury Patients. J Korean Med Sci. 2021 Mar 29;36(12):e80. doi: 10.3346/jkms.2021.36.e80. PMID 33783145